CLINICAL TRIAL: NCT00431184
Title: Effects of Pentazocine Versus Lorazepam on Manic Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Beth L. Murphy MD, PhD, Principal Investigator, Mclean Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006-P-002344
Record Dates: First submitted 2007-02-01; First posted 2007-02-05 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-02

CONDITIONS: Bipolar Disorder; Schizoaffective Disorder; Manic Disorder; Mania; Manic State
Keywords: bipolar disorder; bipolar mania; schizoaffective disorder; schizoaffective mania; mania; kappa opiates; opiates
MeSH Terms: conditions — Bipolar Disorder; Psychotic Disorders; Mania | interventions — Pentazocine; talwin Nx; Lorazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pentazocine then Lorazepam (Active Comparator): In the first leg of the study, pentazocine will be given to subjects randomly assigned to this group. On Day 1, subjects will receive 50mg of pentazocine followed by a second dose of 50mg two hours later. On Day 2, subjects in this group will be given 0.25mg of Lorazepam followed by a second dose of 0.25mg two hours later.
  Interventions: Drug: Pentazocine; Drug: Lorazepam
- Lorazepam then Pentazocine (Active Comparator): In the first leg of the study, lorazepam will be given to subjects randomly assigned to this group. On Day 3, subjects in this group will be given 0.25mg of Lorazepam followed by a second dose of 0.25mg two hours later. On Day 2, subjects will receive 50mg of pentazocine followed by a second dose of 50mg two hours later.
  Interventions: Drug: Pentazocine; Drug: Lorazepam

INTERVENTIONS:
Drug: Pentazocine — see arms description
  Other Names: Talwin Nx
Drug: Lorazepam — see arms description
  Other Names: Ativan

SUMMARY:
Pilot data indicates that pentazocine decreases manic symptoms in hospitalized individuals. To follow up these initial findings, we plan to conduct a larger, more rigorous, double-blind study. We will examine whether pentazocine, an agent with kappa-opiate activity, decreases manic symptoms.

DETAILED DESCRIPTION:
Dysregulation of the opioid system may underlie the pathophysiology of mood disorders, such as bipolar disorder. Drugs that modulate the opioid system might be effective treatments for bipolar disorder. The profile and actions of the kappa-opioid system make drugs that target this system particularly promising as a treatment modality, with relatively low risk of addictive properties. Pentazocine is an approved drug for pain relief with a good side effect profile. It is predominantly a kappa opioid agonist with weaker side effects at mu opioid receptors, at which it is an antagonist. Data from our open-label pilot study of pentazocine had promising results. We will follow up on these findings with a double-blind, active-control study of individuals with bipolar disorder or schizoaffective disorder who are currently hospitalized with acute mania. The antimanic effects of pentazocine will be compared with an active control (ativan).

ELIGIBILITY:
Inclusion Criteria:

* bipolar or schizoaffective disorder
* currently manic
* no acute medical issues
* no substance withdrawal

Exclusion Criteria:

* unable to give informed consent
* using opiates for pain management
* history of head injury, dementia, or mental retardation
* seizure disorder
* glaucoma
* unstable cardiac condition or arrhythmia
* moderate-severe pulmonary disease
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth L Murphy, MD/PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

REFERENCES:
- [Background] Ma J, Ye N, Lange N, Cohen BM. Dynorphinergic GABA neurons are a target of both typical and atypical antipsychotic drugs in the nucleus accumbens shell, central amygdaloid nucleus and thalamic central medial nucleus. Neuroscience. 2003;121(4):991-8. doi: 10.1016/s0306-4522(03)00397-x. PMID 14580949
- [Background] Carlezon WA Jr, Beguin C, DiNieri JA, Baumann MH, Richards MR, Todtenkopf MS, Rothman RB, Ma Z, Lee DY, Cohen BM. Depressive-like effects of the kappa-opioid receptor agonist salvinorin A on behavior and neurochemistry in rats. J Pharmacol Exp Ther. 2006 Jan;316(1):440-7. doi: 10.1124/jpet.105.092304. Epub 2005 Oct 13. PMID 16223871
- [Background] Mague SD, Pliakas AM, Todtenkopf MS, Tomasiewicz HC, Zhang Y, Stevens WC Jr, Jones RM, Portoghese PS, Carlezon WA Jr. Antidepressant-like effects of kappa-opioid receptor antagonists in the forced swim test in rats. J Pharmacol Exp Ther. 2003 Apr;305(1):323-30. doi: 10.1124/jpet.102.046433. PMID 12649385
- [Background] Todtenkopf MS, Marcus JF, Portoghese PS, Carlezon WA Jr. Effects of kappa-opioid receptor ligands on intracranial self-stimulation in rats. Psychopharmacology (Berl). 2004 Apr;172(4):463-70. doi: 10.1007/s00213-003-1680-y. Epub 2004 Jan 16. PMID 14727002
- See also: McLean hospital website, with links to research. — http://www.mclean.harvard.edu

RESULTS

PARTICIPANT FLOW:
Period: 1st Intervention (Day 1)
Arm/Group | Pentazocine Then Lorazepam | Lorazepam Then Pentazocine
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0
Period: Second Intervention (Day 2)
Arm/Group | Pentazocine Then Lorazepam | Lorazepam Then Pentazocine
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pentazocine Then Lorazepam | Lorazepam Then Pentazocine | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Mania Acute Rating Scale (MACS)
Description: Assessment of current mania symptoms using Mania Acute Change Scale (MACS). All 20 questions on the scale have a 0 (absent)-4(most severe) range for describing mania symptoms. The mean MACS score totals were reported, with the total ranging from 0-80. A higher total score indicates a greater number of symptoms and higher symptom intensity, while a smaller score indicates a lesser number of symptoms and higher lower intensity. The change in MACS scores from baseline and those following treatment administration were averaged. The number below represents the average mean change.
Time Frame: On Day 1 and Day 2, at the time of administration of intervention and 5 hours following administration of intervention
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Pentazocine: Subjects received 50mg of pentazocine
- Lorazepam: Subjects received 0.25mg of Lorazepam followed by a second dose of 0.25mg two hours later
Arm/Group | Pentazocine | Lorazepam
Number analyzed (Participants) | 19 | 19
units on a scale | 3.9 [0.7 to 7.1] | 6.4 [3.4 to 9.5]
Statistical Analysis 1: Comparison: Pentazocine vs Lorazepam; Test type: Superiority or Other; p = 0.22, Mixed Models Analysis

2. Secondary Outcome: Young Mania Rating Scale (YMRS)
Description: The YMRS is used to assess manic symptoms. There are 11 questions which ask the patient to rate the severity of symptoms. Scores range from 0 to a maximum of 60. All questions are rated based on severity, with a higher score signifying increased severity. Questions 1-4, 7, and 10 are rated on a 0-4 scale. Questions 5, 6, 8, and 9 are rated on a 0-8 scale.
Time Frame: at the time of administration of intervention and 5 hours following administration of intervention
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Pentazocine: The results below represent the mean change in YMRS scores for all 19 subjects following administration of Pentazocine.
- Lorazepam: The results below represent the mean change in YMRS scores for all 19 subjects following administration of Lorazepam.
Arm/Group | Pentazocine | Lorazepam
Number analyzed (Participants) | 19 | 19
units on a scale | 23.0 [16.6 to 29.4] | 22.6 [15.9 to 29.3]
Statistical Analysis 1: Comparison: Pentazocine vs Lorazepam; Test type: Superiority or Other; p = 0.83, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Data was collected over two contiguous days.
Groups:
- Pentazocine: All subjects receive 50mg of pentazocine followed by a second dose of 50mg two hours later on either Day 1 or Day 2.
- Lorazepam: All subjects receive 0.25mg of Lorazepam followed by a second dose of 0.25mg two hours later on either Day 1 or Day 2.
Arm/Group | Pentazocine | Lorazepam
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No